CLINICAL TRIAL: NCT00447057
Title: A Phase 2 Study of Pemetrexed Versus Pemetrexed Plus Erlotinib in Second-Line Treatment in Patients With Nonsquamous NSCLC
Brief Title: Study of Pemetrexed Versus Pemetrexed Plus Erlotinib as Treatment of Nonsquamous Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10721; H3E-MC-S102 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-09

CONDITIONS: Histological or Cytological Diagnosis of Locally Advanced or Metastatic NSCLC of Nonsquamous Histology and Not Amenable to Curative Therapy.
Keywords: nonsquamous
MeSH Terms: interventions — Pemetrexed; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pemetrexed (Nonsquamous) (Experimental): Group of participants with non-small cell lung cancer (NSCLC) of nonsquamous histology who were assigned to Pemetrexed arm
  Interventions: Drug: Pemetrexed
- Pemetrexed + Erlotinib (Nonsquamous) (Experimental): Group of participants with NSCLC of nonsquamous histology who were assigned to Pemetrexed + Erlotinib arm
  Interventions: Drug: Erlotinib; Drug: Pemetrexed
- Pemetrexed (Squamous) (Experimental): Group of participants with NSCLC of squamous histology who were assigned to Pemetrexed arm
  Interventions: Drug: Pemetrexed
- Pemetrexed + Erlotinib (Squamous) (Experimental): Group of participants with NSCLC of squamous histology who were assigned to Pemetrexed + Erlotinib arm
  Interventions: Drug: Pemetrexed; Drug: Erlotinib

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m² intravenous (iv) over 10 minutes on the first day of each 21-day cycle until disease progression (PD) or unacceptable toxicity
  Other Names: LY231514; Alimta
  Arms: Pemetrexed (Nonsquamous)
Drug: Erlotinib — 150 mg given orally (po), daily (QD), starting on the first day of the first cycle
  Other Names: Tarceva
  Arms: Pemetrexed + Erlotinib (Nonsquamous)
Drug: Pemetrexed — 500 mg/m² iv over 10 minutes on the first day of each 21-day cycle until PD or unacceptable toxicity
  Other Names: LY231514; Alimta
  Arms: Pemetrexed (Squamous); Pemetrexed + Erlotinib (Nonsquamous); Pemetrexed + Erlotinib (Squamous)
Drug: Erlotinib — 150 mg given po, QD, starting on the first day of the first cycle
  Other Names: Tarceva
  Arms: Pemetrexed + Erlotinib (Squamous)

SUMMARY:
This is a multicenter, randomized, Phase 2, open label, parallel trial to evaluate an effect of pemetrexed alone on nonsquamous non-small cell lung cancer (NSCLC) in a second-line setting (such as progression-free survival [PFS], disease control rate, best response rate, time to treatment failure [TTTF], overall survival [OS] and 1-year survival rates) compared to pemetrexed plus erlotinib combination.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of locally advanced or metastatic NSCLC that is of nonsquamous histology and not amenable to curative therapy.
* Failure of previous treatment with one prior platinum-based chemotherapy regimen.
* Good performance status.
* Adequate bone marrow reserve, renal and hepatic functions.

Exclusion Criteria:

* Serious concomitant systemic disease.
* Inability to take oral medication.
* Inability or unwillingness to take vitamin supplementation and corticosteroids.
* Pregnancy / Breast-feeding.
* Treatment with certain medicines that prevent blood from clotting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2007-03; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (23):
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gauting
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gerlingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Immenhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deszk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mátraháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Solna

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 2-arm study; however, results for participant disposition and baseline characteristics are presented for 4 groups including each study arm (Pemetrexed and Pemetrexed + Erlotinib) by histology (Nonsquamous and Squamous). Efficacy results are presented for participants with nonsquamous histology only.
Groups:
- Pemetrexed (Nonsquamous): Pemetrexed: 500 mg/m² intravenous (iv) over 10 minutes on the first day of each 21-day cycle until disease progression or unacceptable toxicity
- Pemetrexed + Erlotinib (Nonsquamous): Pemetrexed: 500 mg/m² iv over 10 minutes on the first day of each 21 day cycle until disease progression or unacceptable toxicity
  Erlotinib: 150 mg given orally (po), daily (QD), starting on the first day of the first cycle
- Pemetrexed (Squamous): Pemetrexed: 500 mg/m² iv over 10 minutes on the first day of each 21 day cycle until disease progression or unacceptable toxicity
- Pemetrexed + Erlotinib (Squamous): Pemetrexed: 500 mg/m² iv over 10 minutes on the first day of each 21 day cycle until disease progression or unacceptable toxicity
  Erlotinib: 150 mg given po, QD, starting on the first day of the first cycle
Period: Overall Study
Arm/Group | Pemetrexed (Nonsquamous) | Pemetrexed + Erlotinib (Nonsquamous) | Pemetrexed (Squamous) | Pemetrexed + Erlotinib (Squamous)
Started | 83 | 76 | 19 | 26
Completed | 0 | 3 | 0 | 0
Not Completed | 83 | 73 | 19 | 26
Not completed — Adverse Event | 4 | 10 | 0 | 3
Not completed — Death due to study disease | 6 | 4 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Entry criteria not met | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 1 | 1
Not completed — Physician Decision | 9 | 6 | 3 | 1
Not completed — Sponsor decision | 1 | 1 | 0 | 0
Not completed — Progressive disease | 58 | 43 | 13 | 18
Not completed — Death due to adverse event | 0 | 0 | 1 | 2
Not completed — Death, study drug related | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed (Nonsquamous): Pemetrexed: 500 mg/m² iv over 10 minutes on the first day of each 21-day cycle until PD or unacceptable toxicity
- Pemetrexed + Erlotinib (Nonsquamous): Pemetrexed: 500 mg/m² iv over 10 minutes on the first day of each 21-day cycle until PD or unacceptable toxicity
  Erlotinib: 150 mg given orally, Daily, starting on the first day of the first cycle
- Pemetrexed (Squamous): Pemetrexed: 500 mg/m² intravenous (iv) over 10 minutes on the first day of each 21 day cycle until disease progression or unacceptable toxicity
- Total: Total of all reporting groups
Arm/Group | Pemetrexed (Nonsquamous) | Pemetrexed + Erlotinib (Nonsquamous) | Pemetrexed (Squamous) | Pemetrexed + Erlotinib (Squamous) | Total
Number analyzed (Participants) | 83 | 76 | 19 | 26 | 204
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.25) | 63.5 (9.70) | 63.9 (9.33) | 66.1 (8.58) | 62.3 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 0 | 2 | 66
  Male | 49 | 46 | 19 | 24 | 138
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 82 | 75 | 19 | 26 | 202
  African | 0 | 0 | 0 | 0 | 0
  Hispanic | 1 | 0 | 0 | 0 | 1
  Native American | 0 | 0 | 0 | 0 | 0
  East Asian | 0 | 0 | 0 | 0 | 0
  West Asian | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Austria | 4 | 5 | 2 | 0 | 11
  Germany | 44 | 37 | 6 | 15 | 102
  Spain | 18 | 9 | 7 | 7 | 41
  Hungary | 12 | 14 | 4 | 4 | 34
  Sweden | 5 | 11 | 0 | 0 | 16
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  0 - Fully Active
  1. - Ambulatory, Restricted Strenuous Activity
  2. - Ambulatory, No Work Activities
  3. - Partially Confined to Bed, Limited Self Care
  4. - Completely Disabled
  Participants
    Status 0 | 33 | 33 | 7 | 9 | 82
    Status 1 | 39 | 33 | 7 | 13 | 92
    Status 2 | 11 | 9 | 5 | 4 | 29
    Unknown | 0 | 1 | 0 | 0 | 1
Basis for Diagnosis [Number; unit: participants]
  Histopathological | 64 | 61 | 18 | 22 | 165
  Cytological | 19 | 15 | 1 | 4 | 39
Initial Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma of the lung | 70 | 61 | 0 | 0 | 131
  Mixed cell (squamous/adenocarcinoma) | 1 | 1 | 0 | 0 | 2
  Large cell lung carcinoma | 6 | 9 | 0 | 0 | 15
  Bronchioalveolar carcinoma | 4 | 1 | 0 | 0 | 5
  Squamous cell carcinoma of the lung | 0 | 0 | 19 | 26 | 45
  Unknown | 2 | 4 | 0 | 0 | 6
Stage of Disease at Study Entry [Number; unit: participants] — Disease Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body).
  Stage 0 - the cancer has not spread beyond the inner lining of the lung Stage I - the cancer is small and hasn't spread to the lymph nodes Stage II - the cancer has spread to some lymph nodes near the original tumor Stage III - the cancer has spread to nearby tissue or spread to far away lymph nodes Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver
  participants
    Stage I | 0 | 0 | 0 | 0 | 0
    Stage II | 0 | 0 | 0 | 0 | 0
    Stage IIIA | 3 | 1 | 2 | 0 | 6
    Stage IIIB | 10 | 11 | 4 | 5 | 30
    Stage IV | 70 | 64 | 13 | 21 | 168
Smoking status [Number; unit: participants]
  Never smoked | 14 | 10 | 0 | 0 | 24
  Ex-smoker | 44 | 51 | 12 | 19 | 126
  Current smoker | 25 | 15 | 7 | 7 | 54
Pack-years, smokers only [Number; unit: participants] — Pack-year equals the number of cigarette packs smoked per day multiplied by the number of years the participant has smoked. For example, 1 pack-year is equal to smoking an average of 20 cigarettes per day (1 pack) for 1 year.
  participants
    Up to 15 pack-years | 5 | 13 | 1 | 1 | 20
    More than 15 pack-years | 60 | 48 | 15 | 25 | 148
    Unknown | 18 | 15 | 3 | 0 | 36

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS per Response Evaluation Criteria in Solid Tumors (RECIST) 1.0 criteria using computed tomography (CT) or magnetic resonance imaging (MRI) for objective determination of progressive disease (PD: ≤20% increase in sum of longest diameter of target lesion). For participants alive as of data cut-off date who did not have PD, PFS was censored at date of last CT/MRI. For participants who received subsequent systemic anticancer therapy (after study discontinuation) prior to PD or death, PFS censored at date of last CT/MRI prior to initiation of post discontinuation systemic anticancer therapy.
Time Frame: Baseline to date of measured PD or death from any cause. Maximum follow-up was from baseline to 32.2 months
Population: Includes Nonsquamous population only.
  In Pemetrexed arm, 13 (15.7%) participants censored overall: 12 (14.5%) because of receiving subsequent systemic anticancer therapy.
  In Pemetrexed + Erlotinib arm, 16 (21.1%) participants censored overall: 9 (11.8%) because of receiving subsequent systemic anticancer therapy.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pemetrexed (Nonsquamous): Pemetrexed: 500 mg/m² intravenous (iv) over 10 minutes on the first day of each 21 day cycle until disease progression or unacceptable toxicity
- Pemetrexed + Erlotinib (Nonsquamous): Pemetrexed: 500 mg/m² intravenous (iv) over 10 minutes on the first day of each 21 day cycle until disease progression or unacceptable toxicity
  Erlotinib: 150 mg given orally, Daily, starting on the first day of the first cycle
Arm/Group | Pemetrexed (Nonsquamous) | Pemetrexed + Erlotinib (Nonsquamous)
Number analyzed (Participants) | 70 | 60
months | 2.9 [1.94 to 3.38] | 3.2 [2.86 to 4.70]
Statistical Analysis 1: Comparison: Pemetrexed (Nonsquamous) vs Pemetrexed + Erlotinib (Nonsquamous); Test type: Superiority or Other; p = 0.0047, Log Rank; Log-rank test with 1-sided alpha of 0.20; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.438 to 0.897]

2. Secondary Outcome: Percentage of Participants With Best Response of Stable Disease (SD), Partial Response (PR) or Complete Response (CR) (Disease Control Rate)
Description: Per RECIST:
  CR: Disappearance of all target lesions; PR: Either a) ≤30% decrease in sum of longest diameter (LD) of target lesions or b) complete disappearance of target lesions, with persistence (but not worsening) of ≥1 nontarget lesions. In either case, no new lesions may have appeared.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
  PD: ≤20% increase in sum of LD of target lesions. Disease Control Rate (%) = (SD+PR+CR)/number of participants in arm*100.
Time Frame: Baseline to measured PD. Maximum follow-up was from Baseline to 34 months
Population: Includes nonsquamous population only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed (Nonsquamous) | Pemetrexed + Erlotinib (Nonsquamous)
Number analyzed (Participants) | 83 | 76
percentage of participants | 51.8 [40.6 to 62.9] | 55.3 [43.4 to 66.7]
Statistical Analysis 1: Comparison: Pemetrexed (Nonsquamous) vs Pemetrexed + Erlotinib (Nonsquamous); Test type: Superiority or Other; p = 0.3909, Fisher Exact

3. Secondary Outcome: Percentage of Participants With Best Response of Complete Response (CR) or Partial Response (PR) (Response Rate)
Description: CR: Disappearance of all tumor lesions; PR: Either a) at least a 30% decrease in sum of LD of target lesions or b) complete disappearance of target lesions, with persistence (but not worsening) ≥1 nontarget lesions. In either case, no new lesions may have appeared.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
  PD: ≤20% increase in the sum of LD of target lesions. Response Rate (%) = (CR+PR)/number of participants in arm*100.
Time Frame: Baseline to measured progressive disease. Maximum follow-up was from Baseline to 34 months
Population: Includes nonsquamous population only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed (Nonsquamous) | Pemetrexed + Erlotinib (Nonsquamous)
Number analyzed (Participants) | 83 | 76
percentage of participants | 10.8 [5.1 to 19.6] | 17.1 [9.4 to 27.5]
Statistical Analysis 1: Comparison: Pemetrexed (Nonsquamous) vs Pemetrexed + Erlotinib (Nonsquamous); Test type: Superiority or Other; p = 0.1808, Fisher Exact

4. Secondary Outcome: Time to Treatment Failure (TTTF)
Description: Defined as the time from randomization to death from any cause, first observation of PD, or study treatment discontinuation due to any reason other than "protocol complete" or "satisfactory response". For participants who discontinued due to "protocol complete" or "satisfactory response", or for participants not known to have discontinued as of the data cut-off date, TTTF was censored at the last contact date.
Time Frame: Baseline to first date among death from any cause, PD, or study treatment discontinuation for any reason other than "protocol complete" or "satisfactory response". Maximum follow-up was from Baseline to 32.2 months
Population: Includes nonsquamous population only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed (Nonsquamous) | Pemetrexed + Erlotinib (Nonsquamous)
Number analyzed (Participants) | 83 | 73
months | 2.4 [1.74 to 2.99] | 3.0 [2.23 to 4.07]
Statistical Analysis 1: Comparison: Pemetrexed (Nonsquamous) vs Pemetrexed + Erlotinib (Nonsquamous); Test type: Superiority or Other; p = 0.0034, Log Rank — 1-sided significance level of 0.20; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.457 to 0.887]

5. Secondary Outcome: Overall Survival (OS)
Description: OS time is the duration from randomization to the date of death from any cause. For each participant who was not known to have died as of the data inclusion cut-off date, OS was censored at the date of last contact.
Time Frame: Baseline to date of death from any cause. Maximum follow-up was from Baseline to 42.6 months.
Population: Pemetrexed arm: 17 (20.5%) participants censored Pemetrexed + Erlotinib arm: 28 (36.8%) participants censored
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed (Nonsquamous) | Pemetrexed + Erlotinib (Nonsquamous)
Number analyzed (Participants) | 66 | 48
months | 7.8 [5.29 to 10.41] | 11.8 [8.18 to 16.66]
Statistical Analysis 1: Comparison: Pemetrexed (Nonsquamous) vs Pemetrexed + Erlotinib (Nonsquamous); Test type: Superiority or Other; p = 0.0190, Log Rank — 1-sided significance level of 0.20; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.465 to 0.981]

6. Secondary Outcome: Percentage of Participants Surviving at 1 Year
Description: Overall Survival (OS) rate at 1 year from the date of randomization was determined using the distribution of OS times and was estimated using the Kaplan-Meier method.
Time Frame: Baseline to date of death from any cause up to 1 year
Population: Includes nonsquamous population only.
  On the Pemetrexed arm, 17 participants were censored overall and on the Pemetrexed + Erlotinib arm, 28 participants were censored overall.
Measure: Median (95% Confidence Interval); unit: Percentage participants with OS ≥1 year
Arm/Group | Pemetrexed (Nonsquamous) | Pemetrexed + Erlotinib (Nonsquamous)
Number analyzed (Participants) | 66 | 48
Percentage participants with OS ≥1 year | 34.1 [23.82 to 44.56] | 49.4 [37.25 to 60.36]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Summaries of serious AEs (SAEs) and all other non-serious AEs are located in the Reported Adverse Event Module.
Time Frame: Baseline up to 42.2 months
Population: All participants who received at least 1 dose of study drug were analyzed for safety. Nonsquamous and squamous populations are combined.
Measure: Number; unit: participants
Groups:
- Pemetrexed (Nonsquamous and Squamous): Pemetrexed: 500 mg/m² intravenous (iv) over 10 minutes on the first day of each 21 day cycle until disease progression or unacceptable toxicity
- Pemetrexed + Erlotinib (Nonsquamous and Squamous): Pemetrexed: 500 mg/m² intravenous (iv) over 10 minutes on the first day of each 21 day cycle until disease progression or unacceptable toxicity
  Erlotinib: 150 mg given orally, Daily, starting on the first day of the first cycle
Arm/Group | Pemetrexed (Nonsquamous and Squamous) | Pemetrexed + Erlotinib (Nonsquamous and Squamous)
Number analyzed (Participants) | 102 | 102
participants
  serious adverse events | 43 | 53
  other adverse events | 91 | 98

ADVERSE EVENTS:
Arm/Group | Pemetrexed (Nonsquamous and Squamous) | Pemetrexed + Erlotinib (Nonsquamous and Squamous)
Serious Adverse Events (participants affected / at risk) | 43/102 | 53/102
Other Adverse Events (participants affected / at risk) | 91/102 | 98/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (Nonsquamous and Squamous) (N=102) | Pemetrexed + Erlotinib (Nonsquamous and Squamous) (N=102)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 10 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 10 (10)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 7 (8)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 2 (2) | 9 (9)
Pain (General disorders) | 2 (2) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (5) | 2 (3)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Candida pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (4) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyothorax (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Superior vena caval occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (Nonsquamous and Squamous) (N=102) | Pemetrexed + Erlotinib (Nonsquamous and Squamous) (N=102)
Anaemia (Blood and lymphatic system disorders) | 22 (26) | 26 (31)
Leukopenia (Blood and lymphatic system disorders) | 9 (20) | 29 (69)
Lymphopenia (Blood and lymphatic system disorders) | 5 (6) | 7 (14)
Neutropenia (Blood and lymphatic system disorders) | 14 (24) | 28 (69)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (9) | 18 (28)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 12 (12) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 44 (60)
Nausea (Gastrointestinal disorders) | 24 (30) | 32 (43)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 13 (14)
Vomiting (Gastrointestinal disorders) | 9 (13) | 15 (19)
Asthenia (General disorders) | 16 (23) | 17 (20)
Chest pain (General disorders) | 6 (6) | 5 (6)
Fatigue (General disorders) | 19 (24) | 22 (27)
Oedema peripheral (General disorders) | 8 (8) | 8 (9)
Pyrexia (General disorders) | 10 (12) | 17 (21)
Nasopharyngitis (Infections and infestations) | 6 (7) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (6) | 17 (21)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 10 (14)
Blood creatinine increased (Investigations) | 5 (7) | 6 (6)
Haemoglobin decreased (Investigations) | 6 (6) | 10 (13)
Weight decreased (Investigations) | 20 (20) | 27 (27)
Decreased appetite (Metabolism and nutrition disorders) | 13 (15) | 31 (33)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7)
Dizziness (Nervous system disorders) | 12 (12) | 12 (12)
Dysgeusia (Nervous system disorders) | 0 (0) | 6 (6)
Headache (Nervous system disorders) | 6 (6) | 6 (6)
Polyneuropathy (Nervous system disorders) | 2 (2) | 9 (9)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 14 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 18 (19)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (10)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 14 (16)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 9 (25) | 43 (48)

LIMITATIONS AND CAVEATS:
Baseline Characteristics are presented by histology (nonsquamous/squamous) for each arm. Per the protocol amendment of August 2008, study entry criteria were changed to exclude participants with predominantly squamous cell histology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days